CLINICAL TRIAL: NCT06199154
Title: Induction of Labor in Morbidly Obese Patients: Comparison of 50 mcg and 25 mcg Misoprostol - A Randomized Control Trial
Brief Title: Induction of Labor in Morbidly Obese Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00108436
Record Dates: First submitted 2023-12-04; First posted 2024-01-10 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Morbid Obesity; Pregnancy
Keywords: induction of labor; morbid obesity; misoprostol
MeSH Terms: conditions — Obesity, Morbid | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control - 25 mcg vaginal misoprostol (Active Comparator): Participants will receive 25 mcg vaginal misoprostol every 4 hours.
  Interventions: Drug: Misoprostol
- Intervention - 50 mcg vaginal misoprostol (Experimental): Participants will receive 50 mcg vaginal misoprostol every 4 hours.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Participants will receive with 25 mcg or 50 mcg vaginal misoprostol every 4 hours.

SUMMARY:
The goal of this randomized control trial is to compare different doses of Misoprostol (25 mcg vs 50 mcg) in induction of labor (IOL) in morbidly obese patients with BMI >40. It is known that morbid obesity is a risk factor for failed IOL and ultimately cesarean delivery (CD.) If the rates of vaginal delivery in this population can improve, then surgical morbidity can be reduced in these patients.

DETAILED DESCRIPTION:
The rate of IOL continues to increase, from about 10% in 1990 to 23% in 2018. Patients with BMI >40 are at increased risk for failed IOL and needing a CD. Studies show that morbidly obese patients require higher doses of pitocin and multiple agents to achieve vaginal delivery, but optimal dosing of misoprostol has not been studied as well. Increasing the rate of vaginal delivery in this population will help decrease risk of surgical morbidity.

The investigators plan to conduct a randomized controlled double blinded trial. Patients who are scheduled for induction of labor after 34 weeks gestation, have a BMI >40, and meet all study inclusion criteria will be approached by research personnel during their outpatient appointments. Participants will be randomized to either receive 25 mcg vaginal misoprostol every 4 hours or 50 mcg vaginal misoprostol every 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese (BMI ≥ 40 kg/m2) at admission for induction of labor
* Speaks English or Spanish
* Gestational age between 34 weeks and 0 days and 42 weeks and 6 days
* Age 18 years old or older
* Viable, single, cephalic fetus
* Intent to proceed with cervical ripening - cervical exam: dilation < 5 cm
* Contractions < 5 per 10 minutes

Exclusion Criteria:

* History of cesarean delivery
* Contraindication to prostaglandin administration (significant myomectomy, prior cesarean delivery)
* Contraindication to vaginal delivery (placenta previa, vasa previa, HIV with high viral load)
* Contraindications to labor (cardiac, neurosurgical, need for cesarean)
* Age < 18yo
* Fetal growth restriction with abnormal umbilical artery Doppler indices
* Cervical dilation >5 cm
* Contractions >5 per 10 minutes
* Significant vaginal bleeding with concern for placental abruption
* Non-reassuring fetal status or fetal heart rate decelerations
* Fetal demise or major fetal anomaly
* Inability to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Achievement of complete cervical dilation | Start of IOL until complete dilation

SECONDARY OUTCOMES:
Time interval from start of induction of labor (IOL) to complete cervical dilation | Start of IOL until complete dilation
Achievement of 6 cm cervical dilation/active labor | Start of IOL until 6 cm dilation
Time interval from start of IOL to 6 cm cervical dilation/active labor | Start of IOL until 6 cm dilation
Time interval from start of IOL to vaginal delivery | Start of IOL until delivery
Time interval from start of IOL to delivery | Start of IOL until delivery
Incidence of vaginal deliveries | Start of IOL until delivery
Incidence of cesarean deliveries | Start of IOL until delivery
Indication for cesarean delivery | Start of IOL until delivery
  Maternal or Fetal
Cervical exam at time of cesarean delivery | Start of IOL until delivery
Number of patients with tachysystole | Start of IOL until delivery
Number of patients with tachysystole with non reassuring fetal heart rate (NRFHT) | Start of IOL until delivery
Number of patients requiring terbutaline | Start of IOL until delivery
Number of patients with chorioamnionitis | Start of IOL until delivery
Number of patients with postpartum hemorrhage | Start of IOL until discharge, assessed up to 4 days
Composite maternal morbidity (need for transfusion, sepsis, ICU admission, death) | Start of IOL until postpartum day 4
Composite neonatal morbidity (NICU admission, Apgar score =<7 at 5 minutes, sepsis, cord gas arterial pH <7.10 and/or base deficit < -12, active cooling protocol, death) | Start of IOL until discharge or day of life 30

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoyert, Donna L. "Maternal Mortality Rates in the United States, 2021." Centers for Disease Control and Prevention, Centers for Disease Control and Prevention, 16 Mar. 2023, www.cdc.gov/nchs/data/hestat/maternal-mortality/2021/maternal-mortality-rates-2021.htm.
- [Background] MarchofDimes. "Total Cesarean Deliveries by Maternal Race/Ethnicity: United States, 2019-2021 Average." March of Dimes | PeriStats, www.marchofdimes.org/peristats/data?reg=99&top=8&stop=356&lev=1&slev=1&obj=1. Accessed 14 Nov. 2023.
- [Background] "Adult Obesity Facts." Centers for Disease Control and Prevention, Centers for Disease Control and Prevention, 17 May 2022, www.cdc.gov/obesity/data/adult.html.
- [Background] Ellis JA, Brown CM, Barger B, Carlson NS. Influence of Maternal Obesity on Labor Induction: A Systematic Review and Meta-Analysis. J Midwifery Womens Health. 2019 Jan;64(1):55-67. doi: 10.1111/jmwh.12935. Epub 2019 Jan 16. PMID 30648804
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Beckwith L, Magner K, Kritzer S, Warshak CR. Prostaglandin versus mechanical dilation and the effect of maternal obesity on failure to achieve active labor: a cohort study. J Matern Fetal Neonatal Med. 2017 Jul;30(13):1621-1626. doi: 10.1080/14767058.2016.1220523. Epub 2016 Aug 25. PMID 27560557
- [Background] O'Dwyer V, O'Kelly S, Monaghan B, Rowan A, Farah N, Turner MJ. Maternal obesity and induction of labor. Acta Obstet Gynecol Scand. 2013 Dec;92(12):1414-8. doi: 10.1111/aogs.12263. PMID 24116732
- [Background] Pevzner L, Powers BL, Rayburn WF, Rumney P, Wing DA. Effects of maternal obesity on duration and outcomes of prostaglandin cervical ripening and labor induction. Obstet Gynecol. 2009 Dec;114(6):1315-1321. doi: 10.1097/AOG.0b013e3181bfb39f. PMID 19935035
- [Background] Drummond R, Patel M, Myers M, Ritter A, Hurvitz JA, Goetzinger KR, Crimmins SD. Class III obesity is an independent risk factor for unsuccessful induction of labor. AJOG Glob Rep. 2022 Sep 23;2(4):100109. doi: 10.1016/j.xagr.2022.100109. eCollection 2022 Nov. PMID 36311296